CLINICAL TRIAL: NCT02639897
Title: Evaluation of Functional Dimensions of Macintosh Blade During Laryngoscopy in Patients With Normal Mouth Opening: Development of a Feasibility Model for Facilitation of Laryngoscopy in Cases of Mouth Opening Restriction Due to Submucous Fibrosis
Brief Title: Evaluation of Functional Dimensions of Macintosh Laryngoscope Blade During Direct Laryngoscopy in Patients With Normal Mouth Opening
Status: Not yet recruiting | Type: Observational
Sponsor: Sir Ganga Ram Hospital (Other)
Responsible Party: Principal Investigator, Nitin Sethi, DNB, Consultant, Sir Ganga Ram Hospital
Other Study IDs: EC/10/15/901
Record Dates: First submitted 2015-12-13; First posted 2015-12-28 (Estimated); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Submucous Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Direct Laryngoscopy — Tracheal intubation with direct laryngoscopy using Macintosh laryngoscope blade

SUMMARY:
Direct laryngoscopy and intubation is an essential initial aspect of airway access during general anesthesia. To perform the procedure effectively, it requires adequate mouth opening, head and neck movement, and a normal temporo-mandibular joint mobility. Any issue with the above three results in a compromised upper airway at the outset and the condition is known as anticipated difficult airway, i.e. an airway that is difficult to access with conventional laryngoscopy and intubation methods. To overcome the difficulty, either one has to resort to newer advanced technique and equipment or the available conventional technique needs to be refined and modified to suit the requirement. While the former requires extraordinary expertise and finances, an option difficult to achieve in developing countries; the latter warrants focused interest to develop alternative approach with the same set of equipments.

Since submucous fibrosis and the associated restricted mouth opening have taken the proposition of an epidemic owing to widespread use of betel nut and tobacco; these patients, when requiring surgery, are difficult candidates for GA and airway control. The fact that, when they arrive as pre-surgical candidates, they have variable degree of mouth opening restriction, which if approached with a strategy, may be amenable to conventional control of airway. If investigators paint all the patients with mouth restriction as difficult airway, it will result in uncalled surgical, economic, health system and psychological burden. Therefore, it is prudent to undertake research relating to refinement of airway access techniques with the easily available, cheap and user- friendly equipment (conventional laryngoscope), such that a proportion of above stated burden can be reduced.

In view of the above, investigators plan to undertake a study to enhance our working knowledge with a conventional laryngoscope (Macintosh) to facilitate ways to control the airway difficulty secondary to mouth opening restriction. Investigators believe that the prospective knowledge thus generated would help us identify whether there is a feasibility of conventional airway management or an alternative advanced access technique is needed in the first place. This will prevent undue cancellations, delayed surgeries, and patient morbidity.

DETAILED DESCRIPTION:
Upper airway access is one of the essential components of general anaesthesia, and more often than not, it is gained by direct laryngoscopy followed by tracheal intubation. While direct laryngoscopy depends on laryngoscope blade design and the anesthetists' skill set, the ease of tracheal intubation is influenced by the line-of-view to the glottis gained by the laryngoscopy maneuver. In patients with normal mouth opening (≥4.0 cm), the act of conventional airway access is not difficult given that the neck extension and the TMJ joint mobility is within normal limits. Conversely, it becomes difficult in patients who have mouth opening restriction, and hence they are adjudicated as 'anticipated difficult airway' (ADA). The ADA, attracts several issues that, not uncommonly, converges on to time inefficiency, heightened equipment cost, operator anxiety, and unfortunately, patient morbidity. There are many causes of restricted mouth opening, defined technically as reduced inter-incisor distance (IID) including trauma, TMJ movement limitation, intra/extra-oral pathology resulting in pain, or the most common pathology in the Indian subcontinent, oral submucosal fibrosis (SMF). While the pathology itself is a forerunner of oral mitosis, it is the associated restricted mouth opening component that put conventional airway access efforts of the anaesthesiologist in spot, and consequently, a whole, sometimes unnecessary rigmarole has to be activated under the heading of 'advanced approach to ADA'.

Oral submucous fibrosis (SMF) is a well-recognized, potentially malignant progressive condition afflicting the oral cavity that is characterised by a reduced mouth opening. The reduction in mouth opening occurs due a vertical reorientation of collagen fibrils that are normally haphazardly arranged. Of the currently available multiple classifications to identify disease stage/severity, the functional classification based on the inter-incisor distance (IID) seems to be most relevant.

IID forms an important component of airway examination and a value of less than 3-cm is suggestive of difficulty in airway management. However, despite the above, SMF is largely unrecognized as a cause of airway difficulty, and even when recognized, no set protocol is available to ensure (as far as possible) a favourable outcome in terms of least morbidity to the patient, and stress to the anaesthesiology team in question.

Need Assessment for the Study Generally, in a tertiary level centre, with all facilities at hand, cases with a reduced IID are normally tackled using a fiberoptic bronchoscope guided tracheal intubation. However, in India, the burden of this disease lies to a great extent in rural/suburban settings where access to a fiberoptic bronchoscope is unlikely. As a result these cases are referred to 'higher' centres for management. This imposes undue burden (logistics/ financial) onto patients and their families. Hence, there is a great need for anaesthesiologists working at the primary/secondary level healthcare set up to get oriented to this problem and be able to manage it with conventional options (direct laryngoscopy & intubation) available to them.

Scientific Contention Direct laryngoscopy remains the foremost among the various techniques available to access the upper airway and the Macintosh blade has been the most preferred blade type. In order to improve direct laryngoscopy, many modifications of blade design have been tested/ compared with the Macintosh blade, but apparently, the clarity as to which laryngoscope blade is most suited for a given airway remains low. For the majority of practicing anaesthesiologists, the availability of different laryngoscope designs has only increased the hit-and-trial option for laryngoscopy.

Since the time it was first introduced, the Macintosh blade (size 1, 2, 3, 4, and 5) has weathered many newer laryngoscope blade designs and stood by our side with consistent/optimal performance. Per se, from a technical standpoint, although shaped the same, various sizes of the Macintosh blade are not exactly similar, the discrepancy becomes obvious when comparing sizes 1, 2 with 3 & 4. Unfortunately, investigators are still unclear as to how design characteristics and the various sizes of the Macintosh blade impact the process of direct laryngoscopy. Generally, the selection of laryngoscope blade (type and sizes) is largely a function of individual experience and preferences. The absence of predefined parameters for the selection of the most appropriate laryngoscope blade for a given airway remains arbitrary. Apparently, an anaesthesiologist will be able to intubate an adult trachea with any of the laryngoscope blade, however, blade type and size selection assumes significance in the presence of a difficult airway.

The three factors which influence successful direct laryngoscopy performance are:

i) The ability to place the laryngoscope blade tip in vallecular recess and engage the hyoid bone. This requires an adequate length of the blade to be introduced orally to reach the vallecula (transition space between base of the tongue and the epiglottis) position.

ii) The ability to displace the tongue aside for clear view to the glottic-epiglottic region iii) Achieving a clear line-of-sight to the glottis-opening. To ensure that the tip of the laryngoscope blade engages the hyoid by placement in the vallecula, an adequate blade length must be inserted into the oral cavity. Normally, this is easily achieved. However, when faced with a situation involving reduced mouth opening/inter-incisor distance (e.g.as in case of SMF), the length of blade that can be inserted into the oral cavity (functional length) becomes a function of the width of the blade's flange at the incisor point. Thus the size of the flange, corresponding to the width of the blade that must be accommodated in the oral cavity assumes particular significance in patients with reduced inter-incisor gap. Typically, for the Macintosh blade's curved design confers different length to its flange's glossal (concave) and the palatal (convex) surface, the functional width of its flange increases from the tip towards the heel [Figure]. Based on the degree of mouth opening restriction and the available IID (in cm), during preoperative evaluation, one can predict and plan how long a Macintosh blade length will be required and what size of the blade would suffice to be placed orally through the available IID.

Hypothesis Development Marks et al, utilized an x-ray based method to devise a method to evaluate laryngoscope blade design during active laryngoscopy procedure. Technically, they found that Macintosh sizes 3 and 4 have a more refined blade design that provides greater degree of forward space enhancement (FSE, allows greater mandibular space for the tongue to be moved into) than other conventional blades (Miller, Soper, etc.). This FSE-effect gets further magnified with increase in functional length of the blade (the length of the blade inside the oral cavity during active laryngoscopy).

Their elaborate work addressed the performance of the laryngoscope blade (size, type) selection in a theoretical setting. The information gleaned from their assessment offered valuable suggestions on optimal blade position during direct laryngoscopy and included:

i) Mandibular space 'encroachment/enhancement' with the use of different blade types/sizes, and ii) 'Line-of-vision' (view to the glottis) versus 'mandibular space restriction' (space for tongue displacement during laryngoscopy).

However, still, the clinical feasibility of knowledge thus gained from performance assessment facilitated by x-ray/fluoroscopy is difficult to translate into routine clinical practice.

As the investigator prepares to take the conventional direct laryngoscopy process into difficult airway situations where the primary difficulty is due to reduced mouth opening, there is a need to convert theoretical knowledge into clinical suggestions. Investigators thus contend that unless they get accustomed with greater clarity on the use of routine equipments, and analyse their practical feasibility in difficult situations, the element of randomness and subjectivity will continue to be a setback.

ELIGIBILITY:
Inclusion Criteria:

1. Consenting adults
2. Both gender
3. Age: 20-65 years
4. Normal preoperative upper airway evaluation and without the presence of anticipated airway access difficulty
5. Patients scheduled for surgery under general anaesthesia with airway control by direct laryngoscopy and tracheal intubation

Exclusion Criteria:

1. Patient refusal
2. Anticipated airway access difficulty
3. Edentulous patients
4. Patients with dental problem (missing tooth, overlap, cosmetic treatment)
5. Vulnerable Patients: High risk situation, major surgery, extremes of age, obstetric patients
6. Previously difficult airway

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for surgery under general anaesthesia with airway control by direct laryngoscopy and tracheal intubation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-10 (Estimated); Primary Completion 2030-06 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Macintosh Blade Length Measurement (in centimeters) | 0 to 5-minutes
  Length of Macintosh blade size 3 and 4 as such (static) and during active direct laryngoscopy (active).
Macintosh Blade Width Measurement (in centimeters) | 0 to 5-minutes
  Width of Macintosh blade size 3 and 4 as such (static) and during active direct laryngoscopy (active).
Inter-incisor Angle on Macintosh Blade Contact Point (in degrees) | 0 to 5-minutes
  The angle formed by the line between the two contact points, viz. a point formed by upper incisor contact of upper flange curve (convex) of the Macintosh laryngoscope blade, and a point of contact between the lower incisor contact with lower flange curve (concave curve) of the Macintosh laryngoscope blade. The line formed by joining these two contact points with the baseline of the laryngoscope will form an angle. This angle will be noted as functional separation of eugnathic, retrognathic or prognathic maxilo-mandibular orientation

SECONDARY OUTCOMES:
Upper Airway Measurements (in centimeters) | 0 to 5-minutes
  Mento-hyoid, mento-thyroid distance, and the length of sub-mandibular triangle perpendicular
Correlation Assessment | 0 to 5-minutes
  The functional laryngoscope length will be tested for correlation with the linear neck (Mento-hyoid distance, menlo-thyroid distance ) and mandibular distances (perpendicular to sub-mandibular triangle) and the most consistent one will be taken

CONTACTS AND LOCATIONS:
Overall Officials: Amitabh Dutta, MD, Study Director — Sir Ganga Ram Hospital, New Delhi, INDIA; Ameya Pappu, MBBS, Study Chair — Sir Ganga Ram Hospital, New Delhi, INDIA; Nitin Sethi, DNB, Principal Investigator — Sir Ganga Ram Hospital, New Delhi, INDIA
Locations (1):
- Sir Ganga Ram Hospital, New Delhi, India